CLINICAL TRIAL: NCT02167633
Title: A Randomized Trial of Stereotactic Radiosurgery Versus Decompressive Surgery Followed by Postoperative Radiotherapy in Metastatic Spinal Cord Compression
Brief Title: Stereotactic Radiosurgery in Metastatic Spinal Cord Compression
Acronym: Stereocord
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low accrual rate
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Morten Hiul Suppli, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2014-050; RH SRS in MESCC 2014 (Other: Rigshospitalet)
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Compression; Neoplasm Metastasis
Keywords: Radiosurgery; Laminectomy; Radiotherapy; Spinal Cord Compression; Neoplasm Metastasis; Randomized Controlled Trial
MeSH Terms: conditions — Spinal Cord Compression; Neoplasm Metastasis | interventions — Laminectomy; Radiosurgery; Glucocorticoids; Steroids; Pantoprazole; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Decompression surgery plus fractionated radiotherapy (Active Comparator)
  Interventions: Procedure: Decompression surgery; Radiation: Fractionated Radiotherapy; Drug: Glucocorticoids; Drug: Pantoprazole
- Radiosurgery (Experimental): Patients treated with radiosurgery/SBRT will receive a prescribed dose of 16 Gy in one fraction to cover as large a fraction as possible the defined target volume
  Interventions: Radiation: Radiosurgery; Drug: Glucocorticoids; Drug: Pantoprazole

INTERVENTIONS:
Procedure: Decompression surgery — Patients will undergo posterior decompression/laminectomy on relevant spinal levels depending on neurological symptoms. If there is a need of spinal stabilization after decompression, patients will undergo posterior instrumentation with pedicle screws and titanium rods. Instrumentation will be done two or three levels above and below each level with metastatic affection.
  Other Names: laminectomy
  Arms: Decompression surgery plus fractionated radiotherapy
Radiation: Radiosurgery — Patients treated with radiosurgery/SBRT will receive a prescribed dose of 16 Gy in 1 fraction to cover as large a fraction as possible the defined target volume
  Other Names: Stereotactic Body Radiotherapy
  Arms: Radiosurgery
Radiation: Fractionated Radiotherapy — Patients allocated to surgery will receive postoperative radiotherapy commencing between 10 to 21 days after decompressive surgery. Target should include the entire vertebral body and the vertebral arch at the operated level of the vertebral column.
  Patients receiving postoperative radiotherapy will receive 30 Gy in 10 fractions with 3 Gy pr. fraction. The prescribed dose should cover at least 90 % of the defined target volume.
  Arms: Decompression surgery plus fractionated radiotherapy
Drug: Glucocorticoids — All patients referred with clinical suspicion of metastatic spinal cord compression will receive high dose glucocorticoids. Dose adjusted to risc of side effects.
  Other Names: steroids
Drug: Pantoprazole — All patients receiving high dose glucocorticoids will also be prescribed with pantoprazole 40/daily to prevent gastric ulcers
  Other Names: Proton pump inhibitor (PPI)

SUMMARY:
To determine whether stereotactic radiosurgery of metastatic spinal cord compression is equivalent to decompressive surgery followed by external body radiation therapy to maintain ability to walk at 6 weeks.

DETAILED DESCRIPTION:
Metastatic spinal cord compression (MSCC) is an acute event demanding treatment which otherwise would eventually lead to paraplegia in all patients. This is a serious condition for the individual cancer patient and burdensome for the healthcare system. A surgical intervention plus fractionated radiation therapy (FRT) is currently the standard treatment.

Proposed Solution: If spinal cord dose is respected, local tumor control could be equivalent using stereotactic body radiation therapy (SBRT) with minimal risk in comparison to decompression surgery and postoperative conventional radiotherapy without the additional burden on the patient of performing an invasive surgical procedure.

Clinical Impact:

Patients currently requiring surgery plus radiation therapy will potentially benefit form the proposed method. Patients will potentially benefit from reduced toxicity by avoiding the surgical procedure. In addition, a shorter treatment protocol with only one fraction is beneficial.

Aims:

The investigators' hypothesis is that stereotactic body radiation therapy (SBRT) could be equivalent alternative in the case of patients presenting with metastatic spinal cord compression with minor neurologic deficits.

Specific aims:

1. Determine the feasibility of recruiting patients to be randomized towards SBRT vs. of surgery plus FRT
2. Determine the ability to walk after 6 weeks measured from the starting date of treatment
3. Determine the side-effects and quality of life metrics following both treatment arms
4. Determine the rate of local control following therapy using MRI scan

Project Plan:

The investigators intend to investigate if stereotactic body radiation therapy (SBRT) could be equivalent alternative in the case of patients presenting with metastatic spinal cord compression with minor neurologic deficits

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological confirmed malignancy that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective
* Patients must have localized spine metastasis from first cervical to last lumbar vertebra with evidence of radiological SCC (rSCC) on a diagnostic MRI defined as involvement or compression of either the spinal cord or the cauda equina by an epidural mass lesion or metastatic disease causing impingement, indentation or loss of definition of the thecal sac
* A maximum of two separate sites requiring treatment is allowed with maximum two vertebra pr. site
* Eligible for surgery defined by technical assessment by surgeon whether surgical decompression is possible with proper stabilization of the spine
* No medical co-morbidity contradicting anesthesia
* Patient without former treatment for metastatic spinal cord compression with either decompressive surgery and/or radiation therapy
* Patient with mild to moderate neurologic signs are eligible. These neurological signs include radiculopathy, dermatomal sensory change, and muscle strength of involved extremity 4/5 on MRC scale
* Age ≥18 years
* ECOG performance status ≤2
* Life expectancy of greater than 3 months
* The effects of ionizing radiation on the developing human fetus are known to be teratogenic. For this reason women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of radiation therapy administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Histology of myeloma or lymphoma
* Patients with any spine metastasis that is not planned to be treated per protocol
* Spine instability due to a compression fracture or impending vertebral compression fracture
* Patients with rapid neurologic decline within 24 hours
* Bony retropulsion causing neurologic abnormality
* Prior radiation to the index spine
* Patients for whom an MRI of the spine is medically contraindicated
* Patients allergic to contrast dye used in MRIs
* Patients who are receiving any other investigational agents
* Patients with more than two known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patient with any serious neurologic condition other than MSCC that could confound the diagnosis and interpretation of radiation induced myelopathy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Ability to walk | 6 weeks
  Ability to walk determined by EQ-5D-5L

SECONDARY OUTCOMES:
Self reported pain | 0, 6, 12, 26, 52 weeks
  self reported pain determined by EQ-5D-5L
Self reported bladder control | 0, 6, 12, 26, 52 weeks
  reported by questionnaire
Quality of life | 0, 6, 12, 26, 52
  QOL determined by EQ-5D-5L
Response rate | 6 weeks
  Post interventional MRI scan with response classified according to RECIST 1.1
Toxicity and interventional related complications | 0, 6, 12, 26, 52 weeks
  Determined by CTCAE 4.0

OTHER OUTCOMES:
Days of treatment | 52 weeks
  measurement of therapy related treatment days both as ambulatory and admitted to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Morten H Suppli, MD, Principal Investigator — Rigshospitalet, Denmark; Svend Aage Engelholm, MD, Study Director — Rigshospitalet, Denmark; Benny Dahl, MD, Study Chair — Rigshospitalet, Denmark; Helle Pappot, MD, Study Chair — Rigshospitalet, Denmark; Per Munck af Rosenschöld, Medical Physicist, Study Chair — Rigshospitalet, Denmark; Søren S Morgen, MD, Study Chair — Rigshospitalet, Denmark; Ivan Vogelius, Medicial Physicist, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Morgen SS, Lund-Andersen C, Larsen CF, Engelholm SA, Dahl B. Prognosis in patients with symptomatic metastatic spinal cord compression: survival in different cancer diagnosis in a cohort of 2321 patients. Spine (Phila Pa 1976). 2013 Jul 15;38(16):1362-7. doi: 10.1097/BRS.0b013e318294835b. PMID 23574811
- [Background] Patchell RA, Tibbs PA, Regine WF, Payne R, Saris S, Kryscio RJ, Mohiuddin M, Young B. Direct decompressive surgical resection in the treatment of spinal cord compression caused by metastatic cancer: a randomised trial. Lancet. 2005 Aug 20-26;366(9486):643-8. doi: 10.1016/S0140-6736(05)66954-1. PMID 16112300
- [Background] Rades D, Huttenlocher S, Dunst J, Bajrovic A, Karstens JH, Rudat V, Schild SE. Matched pair analysis comparing surgery followed by radiotherapy and radiotherapy alone for metastatic spinal cord compression. J Clin Oncol. 2010 Aug 1;28(22):3597-604. doi: 10.1200/JCO.2010.28.5635. Epub 2010 Jul 6. PMID 20606090
- [Background] George R, Jeba J, Ramkumar G, Chacko AG, Leng M, Tharyan P. Interventions for the treatment of metastatic extradural spinal cord compression in adults. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD006716. doi: 10.1002/14651858.CD006716.pub2. PMID 18843728
- [Background] Rock JP, Ryu S, Yin FF, Schreiber F, Abdulhak M. The evolving role of stereotactic radiosurgery and stereotactic radiation therapy for patients with spine tumors. J Neurooncol. 2004 Aug-Sep;69(1-3):319-34. doi: 10.1023/b:neon.0000041890.01837.53. PMID 15527098
- [Background] Gerszten PC, Burton SA, Ozhasoglu C, Welch WC. Radiosurgery for spinal metastases: clinical experience in 500 cases from a single institution. Spine (Phila Pa 1976). 2007 Jan 15;32(2):193-9. doi: 10.1097/01.brs.0000251863.76595.a2. PMID 17224814
- [Background] Ryu S, Rock J, Jain R, Lu M, Anderson J, Jin JY, Rosenblum M, Movsas B, Kim JH. Radiosurgical decompression of metastatic epidural compression. Cancer. 2010 May 1;116(9):2250-7. doi: 10.1002/cncr.24993. PMID 20209611
- [Background] Jin R, Rock J, Jin JY, Janakiraman N, Kim JH, Movsas B, Ryu S. Single fraction spine radiosurgery for myeloma epidural spinal cord compression. J Exp Ther Oncol. 2009;8(1):35-41. PMID 19827269
- [Background] Sahgal A, Ma L, Gibbs I, Gerszten PC, Ryu S, Soltys S, Weinberg V, Wong S, Chang E, Fowler J, Larson DA. Spinal cord tolerance for stereotactic body radiotherapy. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):548-53. doi: 10.1016/j.ijrobp.2009.05.023. Epub 2009 Sep 16. PMID 19765914
- [Background] Kirkpatrick JP, van der Kogel AJ, Schultheiss TE. Radiation dose-volume effects in the spinal cord. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S42-9. doi: 10.1016/j.ijrobp.2009.04.095. PMID 20171517
- [Background] Timmerman RD. An overview of hypofractionation and introduction to this issue of seminars in radiation oncology. Semin Radiat Oncol. 2008 Oct;18(4):215-22. doi: 10.1016/j.semradonc.2008.04.001. No abstract available. PMID 18725106
- [Background] Boehling NS, Grosshans DR, Allen PK, McAleer MF, Burton AW, Azeem S, Rhines LD, Chang EL. Vertebral compression fracture risk after stereotactic body radiotherapy for spinal metastases. J Neurosurg Spine. 2012 Apr;16(4):379-86. doi: 10.3171/2011.11.SPINE116. Epub 2012 Jan 6. PMID 22225488
- [Background] Cunha MV, Al-Omair A, Atenafu EG, Masucci GL, Letourneau D, Korol R, Yu E, Howard P, Lochray F, da Costa LB, Fehlings MG, Sahgal A. Vertebral compression fracture (VCF) after spine stereotactic body radiation therapy (SBRT): analysis of predictive factors. Int J Radiat Oncol Biol Phys. 2012 Nov 1;84(3):e343-9. doi: 10.1016/j.ijrobp.2012.04.034. Epub 2012 Jun 1. PMID 22658511
- [Background] Choi D, Morris S, Crockard A, Albert T, Bunger C, Fehlings M, Harrop J, Kawahara N, Martin JA, Massicotte EM, Mazel C, Oner FC, Peul W, Tomita K, Wang M. Assessment of quality of life after surgery for spinal metastases: position statement of the Global Spine Tumour Study Group. World Neurosurg. 2013 Dec;80(6):e175-9. doi: 10.1016/j.wneu.2013.02.054. Epub 2013 Feb 16. PMID 23422266
- [Background] Cox BW, Spratt DE, Lovelock M, Bilsky MH, Lis E, Ryu S, Sheehan J, Gerszten PC, Chang E, Gibbs I, Soltys S, Sahgal A, Deasy J, Flickinger J, Quader M, Mindea S, Yamada Y. International Spine Radiosurgery Consortium consensus guidelines for target volume definition in spinal stereotactic radiosurgery. Int J Radiat Oncol Biol Phys. 2012 Aug 1;83(5):e597-605. doi: 10.1016/j.ijrobp.2012.03.009. Epub 2012 May 19. PMID 22608954
- [Background] Tokuhashi Y, Matsuzaki H, Oda H, Oshima M, Ryu J. A revised scoring system for preoperative evaluation of metastatic spine tumor prognosis. Spine (Phila Pa 1976). 2005 Oct 1;30(19):2186-91. doi: 10.1097/01.brs.0000180401.06919.a5. PMID 16205345
- [Derived] Suppli MH, Munck Af Rosenschold P, Dahl B, Berthelsen AK, Engelholm SA, Pappot H. Premature Termination of a Randomized Controlled Trial on Image-Guided Stereotactic Body Radiotherapy of Metastatic Spinal Cord Compression. Oncologist. 2020 Mar;25(3):210-e422. doi: 10.1634/theoncologist.2019-0672. Epub 2019 Oct 11. PMID 32162821